CLINICAL TRIAL: NCT00253162
Title: The Efficacy And Safety Of Flexible Dose Ranges Of Risperidone Versus Placebo Or Haloperidol In The Treatment Of Manic Episodes Associated With Bipolar I Disorder.
Brief Title: A Study of the Effectiveness and Safety of Risperidone Compared With Placebo in the Treatment of Manic Episodes Associated With Bipolar I Disorder, and the Maintenance of Anti-manic Effectiveness of Risperidone Compared With Haloperidol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006049
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Bipolar Disorders; Manic Disorder
Keywords: risperidone; antipsychotic agents; bipolar disorders; manic episode
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of the study is to assess the effectiveness and safety of risperidone (an antipsychotic medication) compared with placebo after 3 weeks of treatment in patients with bipolar disorder who are experiencing manic episodes. A secondary purpose of the study is to assess the maintenance of risperidone effectiveness versus haloperidol (an antipsychotic medication) after 12 weeks of treatment.

DETAILED DESCRIPTION:
Antipsychotic agents have, for a long time, been used to alleviate the severe behavioral problems associated with manic episodes. Risperidone, widely used in the treatment of schizophrenia, has been shown to be effective in the treatment of manic and mixed episodes associated with bipolar disorders. This is a randomized, double-blind study to evaluate the effectiveness and safety of risperidone compared with placebo after 3 weeks of treatment in patients with bipolar disorder who are experiencing manic episodes. A secondary objective is to estimate the difference between the anti-manic efficacy of risperidone and haloperidol (active comparator) after 12 weeks of treatment. Haloperidol also serves as an internal control for the 3-week treatment period. The study has two 2 phases: an acute period consisting of 3 weeks of double-blind treatment (risperidone, haloperidol, or placebo) followed by a maintenance period consisting of 9 weeks of double-blind treatment (risperidone or haloperidol) or 9 weeks of open-label treatment (risperidone). Patients receive study medication to be taken orally once a day at gradually increasing doses during the first week (risperidone, a range of 1 - 6 mg/day or haloperidol, a range of 2 - 12 mg/day) to achieve optimal effectiveness, while minimizing any intolerance to the drug. Daily treatment continues at the optimal dose through Week 3 of the first phase. After completing the 3-week double-blind period, patients can continue double-blind treatment for an additional 9 weeks at the optimal dose (with placebo patients crossed over to risperidone), or enter the 9-week open-label period of risperidone treatment. Adjustment to achieve an optimal dosage is made for those patients whose medication is changed upon entering the second phase.

The primary measure of effectiveness (acute efficacy) is the change in Young Mania Rating Scale (YMRS) total score from baseline to the endpoint at 3 weeks of the acute treatment period. Additional efficacy measures for the study assess maintenance efficacy. These measures include the Clinical Global Impression-Severity of Illness (CGI-S) scale; Global Assessment Scale (GAS), which assesses the patient's level of functioning; Brief Psychiatric Rating Scale (BPRS), a scale for measuring psychotic symptoms; and the Montgomery Asberg Depression Rating Scale (MADRS), which evaluates symptoms of depression. Safety assessments include the incidence of adverse events and measurement of vital signs (temperature, pulse, blood pressure) throughout the study; evaluation of the presence and severity of extrapyramidal symptoms by the Extrapyramidal Symptom Rating Scale (ESRS) at specified intervals; and clinical laboratory tests (hematology, biochemistry, urinalysis) at the start and end of both phases of the study. The study hypothesis is that 3 weeks of daily treatment with risperidone is more effective than placebo, as measured by Young Mania Rating Scale scores, in the treatment of the manic phase of Bipolar I Disorder. Acute phase: Risperidone orally, once-daily: 2 mg on Day 1, 1 - 3 mg on Days 2 to 4, and 1 - 6 mg on Days 5 to 21; or haloperidol orally, once-daily: 4 mg on Days 1 to 4 and 2 - 12 mg on Days 5 to 21; or placebo orally, once-daily Days 1 to 21. Maintenance phase: optimal dose of risperidone or haloperidol for 9 weeks (placebo patients cross over to risperidone) or Open-label phase: risperidone for 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnosis criteria for Bipolar I Disorder - Most Recent Episode Manic (Diagnostic and Statistical Manual of Mental Diseases, 4th edition, (DSM-IV))
* meets DSM-IV criteria for a current manic episode
* hospitalized voluntarily at study initiation
* history of at least one documented manic or mixed episode prior to study initiation
* total score of >=20 on the Young Mania Rating Scale (YMRS) and total score of <=20 on the Montgomery Asberg Depression Rating Scale (MADRS) at start of the study

Exclusion Criteria:

* Meets DSM-IV criteria for Schizoaffective Disorder or for rapid cycling
* borderline or antisocial personality disorder
* history of substance dependence (excluding nicotine and caffeine) within the 3 months prior to study initiation
* seizure disorder
* females who are pregnant or nursing, or those lacking adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2001-03; Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Acute efficacy: Change in Young Mania Rating Scale (YMRS) total score from baseline to endpoint of 3 weeks of acute treatment period.

SECONDARY OUTCOMES:
Maintenance efficacy: Young Mania Rating Scale, Clinical Global Impression-Severity of Illness scale, Global Assessment Scale, Brief Psychiatric Rating Scale, Montgomery Asberg Depression Rating Scale; incidence of adverse events throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Smulevich AB, Khanna S, Eerdekens M, Karcher K, Kramer M, Grossman F. Acute and continuation risperidone monotherapy in bipolar mania: a 3-week placebo-controlled trial followed by a 9-week double-blind trial of risperidone and haloperidol. Eur Neuropsychopharmacol. 2005 Jan;15(1):75-84. doi: 10.1016/j.euroneuro.2004.06.003. PMID 15572276